CLINICAL TRIAL: NCT06046976
Title: Evaluation of Piezosurgical vs Conventional Surgery Approach During Complex Exodontia in Healthy and Patients With Diabetes Mellitus Type 2
Brief Title: Piezosurgical vs Conventional Exodontia Surgery in Healthy and Patients With Diabetes Mellitus Type 2
Acronym: PCSDMT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Bozidar Brkovic, DDS, MSc, PhD, Professor, DDS PhD, Professor, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 36/06
Record Dates: First submitted 2022-12-02; First posted 2023-09-21 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2; Surgery; Tooth Extraction Status Nos
Keywords: piesosurgery; exodontia; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy (Active Comparator)
  Interventions: Procedure: piesosurgical extraction; Procedure: conventional extraction
- Diabetes mellitus type 2 (Experimental)
  Interventions: Procedure: piesosurgical extraction; Procedure: conventional extraction

INTERVENTIONS:
Procedure: piesosurgical extraction — exodontia of multi - rooted teeth in upper/lower jaw using piesosurgical approach
Procedure: conventional extraction — exodontia of multi - rooted teeth in upper/lower jaw using piesosurgical approach

SUMMARY:
This study will evaluateand compare intraoperative and postoperative clinical parameters related to discomfort and wound heeling, as well as laboratory wound healing parameters after piezosurgical and conventional surgery approach during complex exodontia in healthy and patients with Diabetes Mellitus Type 2

ELIGIBILITY:
Inclusion Criteria:

* multiple multi-rooted teeth indicated for extraction
* controlled DMT2

Exclusion Criteria:

* HbA1c >7%
* chronic orofacial pain and infection in orofacial region
* alcohol and tobacco consumption
* pregnant women and nursing mothers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Duration of osteotomy | from the start of procedure to the end of performing osteotomy
MicroRNA 21 (Mir-21) expression | during the first 24 hours after intervention

SECONDARY OUTCOMES:
Duration of tooth sectioning | from the beginning of tooth sectioning to the end of tooth sectioning
Total exodontia time | from the beginning of surgical procedure to the end of tooth extraction
Pain intensity | during the first 24 hours after intervention
  Numerical Rating Scale, measuring pain intensity ranging from 0 (no pain) to 10 (the worst pain imaginable)
Healing Index Score | within 21 days after procedure
  3 scoring levels for each of the 4 parameters considered: tissue color (1 = 100% of gingiva pink; 2 = <50% of gingiva red, hyper- emic, movable; 3 = >50% of gingiva red, hyperemic, movable), color and consistency of the healing tissue (1 = close grained, pink; 2 = soft, red; 3 = fragile, greenish or grayish), suppuration (1 = absent; 2 = absent but pronounced amount of plaque around socket walls; 3 = pronounced), and bleeding (1 = absent; 2 = induced by palpation; 3 = spontaneous). Thus, the scoring scale ranged from 4, corresponding to excellent healing, to 12, indicating severely impaired healing.
First postoperative pain report | within 24 hours after procedure
  time between the end of procedure and first pain experienced by the patient measured in minutes
First analgesic consumption | within 24 hours after procedure
  time from the end of the procedure until first analgesic consumption measured in minutes
Clinical appearance of gingival tissue | within 7 days after procedure
  clinical appearance of the soft tissues (Visual Analogue Scale 0 to 3, according to the color and presence of edema and bleeding; ie, 0, normally pink, not edematous; 1, pink-red, slightly edematous; 2, red, edematous; and 3, red, edematous, bled easily when touched
Residual Socket Volume | within 21 days after procedure
  the residual socket volume (RSV) is the fraction of the postextraction original cavity still open at each follow-up session (t = 3, 7, 14, and 21 days), computed as the ratio of mesiodistal (MD), bucolingual (BL) and socket depth (SD) at the follow-up session to the baseline value (t=0), measured after extraction (perfect closure corresponds to RSV = 0.00)
Postextraction wound epithelization | within 21 days after procedure
  Epithelialization was measured as bucolingual and mesiodistal diameter of the extraction socket during the follow-up (3, 7, 14 and 21 postoperative day), expressed in millimeters
Vascular Endothelial Growth Factor (VEGF) level | within 24 hours after intervention
  detected by Enzyme-Linked Immunosorbent Essay method
Matrix Metalloproteinase 9 (MMP9) level | within 24 hours after intervention
  detected by Enzyme-Linked Immunosorbent Essay method
Phosphatase and Tensin Homolog (PTEN) level | within 24 hours after intervention
  detected by Enzyme-Linked Immunosorbent Essay method
Superoxide Dismutase(SOD) enzyme activity (%) | within 24 hours after intervention
  Activity level detected by spectrophotometry using SOD Assay kit

CONTACTS AND LOCATIONS:
Overall Officials: Milan Vucetic, DDS PHD, Principal Investigator — University of Belgrade Faculty of Dental Medicine; Bozidar Brkovic, DDS PhD, Study Director — University of Belgrade Faculty of Dental Medicine; Marija S Milic, DDS PhD, Principal Investigator — University of Belgrade Faculty of Dental Medicine; Jelena Roganovic, DDS PhD, Principal Investigator — University of Belgrade Faculty of Dental Medicine
Locations (1):
- University of Belgrade Faculty of Dental Medicine, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP